CLINICAL TRIAL: NCT02755675
Title: uPAR-PET for Prognostication in Patients With Non-small Cell Lung Cancer, Malignant Pleural Mesothelioma and Large Cell Neuroendocrine Carcinoma of the Lung
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Malene Martini Clausen, MD, PhD, postdoc, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AK-2015-LC-1
Record Dates: First submitted 2016-04-19; First posted 2016-04-29 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Non-small Cell Lung Cancer; Malignant Pleural Mesothelioma; Large Cell Neuroendocrine Carcinoma of the Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 68Ga-NOTA-AE105 PET/CT (Experimental): One injection of 68Ga-NOTA-AE105 followed by positron emission tomography/computed tomography (PET/CT scan) will be performed before treatment start to evaluate the prognostic value of uPAR PET/CT.
  Interventions: Other: 68Ga-NOTA-AE105 PET/CT

INTERVENTIONS:
Other: 68Ga-NOTA-AE105 PET/CT — Following injection of 68Ga-NOTA-AE105 the patients will be subjected to PET/CT

SUMMARY:
uPAR PET/CT as a prognostic marker in non-small cell lung cancer.

DETAILED DESCRIPTION:
Study I: uPAR PET/CT with 68Ga-NOTA-AE105 will be evaluated as a prognostic tool in patients with non-small cell lung cancer (NSCLC) (stage IV (Ia) operable disease (Ib)) by observer-blinded readings and compared to the prognostic performance of FDG PET/CT and prognostic biomarkers as uPAR.

Furthermore, uPAR PET/CT will be evaluated in a pilot study in patients with malignant pleural mesothelioma (MPM) (Study II) and large cell neuroendocrine carcinoma of the lung (LCNEC) (Study III) and correlated with immunohistochemical uPAR expression.

ELIGIBILITY:
Inclusion Criteria:

Study I

* Histologically verified NSCLC (Study I)
* Stage IV disease
* Operable disease
* The participants must be capable of understanding and giving full informed written consent

Study II

* Histologically verified MPM (Study II)
* The participants must be capable of understanding and giving full informed written consent

Study III

* Histologically verified LCNEC (Study III)
* The participants must be capable of understanding and giving full informed written consent

Exclusion Criteria:

Study I, II, III

* Pregnancy
* Lactation/breast feeding
* Treatment with neoadjuvant chemotherapy
* Weight above 140 kg
* Allergy to 68Ga-NOTA-AE105

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-04; Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Study Ia: Overall survival (OS) | Study Ia: OS is evaluated after clinical follow-up for 18 months (stage IV disease)
Study Ib: Overall survival (OS) | Study Ib: OS is evaluated after clinical follow-up for 60 months (operable disease)
Study II and III: Uptake of 68Ga-NOTA-AE105 in primary tumor lesion (dichotomized +/-) | Study II and III: Uptake of 68Ga-NOTA-AE105 is evaluated based on PET/CT scans performed within 1 hour post injection of 68Ga-NOTA-AE105

SECONDARY OUTCOMES:
Study Ia: Progression free survival (PFS) | Study Ia: PFS is evaluated after clinical follow-up for 18 months (stage IV disease)
Study Ib: Disease free survival (DFS) | Study Ib: DFS is evaluated after clinical follow-up for 60 months (operable disease)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No